CLINICAL TRIAL: NCT02296294
Title: Body Composition Monitoring for Determination of the Fluid Status in Volunteers Undergoing Intravenous Fluid Therapy
Acronym: BCM_Volunteer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Kabon, MD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: BCM Volunteer Study
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Fluid Shifts; Body Fluid Compartments
Keywords: Bioimpedance Spectroscopy, Body Composition Monitor, Fluid Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluid Therapy (Active Comparator): Intravenous isotonic fluid therapy of Elo-mel® (Fresenius Kabi Austria) at a rate of 0,50ml/kg/min for one hour.
  Body Composition Monitoring every 10 minutes for 6hours.
  Interventions: Drug: Elo-mel® (Fresenius Kabi Austria); Device: Body Composition Monitoring
- Zero Therapy (Placebo Comparator): Body Composition Monitoring every 10 minutes for 6hours. No intravenous fluid therapy
  Interventions: Device: Body Composition Monitoring

INTERVENTIONS:
Drug: Elo-mel® (Fresenius Kabi Austria) — an iv isotonic crystalloid fluid therapy at a rate of 0,50ml/kg/min for one hour.
  Arms: Fluid Therapy
Device: Body Composition Monitoring — BCM measurements every 10 minutes for 6 hours.
  Other Names: BCM

SUMMARY:
This volunteer study tests a recently developed whole-body bioimpedance spectroscopy device called Body Composition Monitor (BCM) which measures the body composition (i.e. the water content of the body).

Specifically, the investigators will evaluate the use of BCM for correct detection of intravenous administered crystalloids in the volunteers´ fluid compartments. Furthermore we will test the change over time of the volunteers´ volume status after an intravenous fluid therapy.

DETAILED DESCRIPTION:
Technically assisted assessment of volume status may be useful to direct fluid administration.

As a prerequisite the investigators will test a recently developed whole-body bioimpedance spectroscopy device to determine fluid status in volunteers after an intravenous fluid therapy.

The correlation of infused fluid and change of the fluid status measured with Body Composition Monitor (BCM, Fresenius Medical Care, Germany) is still unknown.

Using a three-compartment physiologic tissue model, BCM determine total body fluid volume (TBV), extracellular volume (ECV), intracellular volume (ICV) and fluid overload (FO) as surplus or deficit of 'normal' extracellular volume. The BCM device measures resistance and reactance at 50 discrete frequencies covering the frequency spectrum from 5 to 1000 kHz through the entire patient via 4 electrodes placed on the wrist and ankle.

Fifteen volunteers will be enrolled in a randomized, blinded cross over study. After randomisation into one of two treatments the volunteer will receive either an iv isotonic fluid therapy of Elo-mel® (Fresenius Kabi Austria) at a rate of 0,50ml/kg/min for one hour or no fluid therapy. At the second study day the volunteer will obtain the opposite treatment.

We will perform BCM measurements every 10 minutes before, during and after the treatment for 6 hours or until the BCM results return to baseline. The results are stored on a BCM patient card automatically.

The main objective of this study is to detect the administered iv fluid in the extracellular compartment respectively in FO, TBV and ICV.

Secondary outcome parameters include the change over time of ICV, ECV, TBV and FO after the iv therapy at the study day "Fluid Therapy".

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged between 18 and 50 years
* BMI < 30 kg/m2
* Written informed consent given by volunteers after being provided with detailed information about the nature, risks, and scope of the clinical study

Exclusion Criteria:

* Implanted pacemaker or defibrillator
* Limb amputation identified by physical examination
* Known allergy or hypersensitivity to Elo-Mel
* Abnormalities in Blood pressure (Hypotension with a systolic BP < 90 mmHg and hypertension with a systolic BP > 160 mmHg) after 5 min resting
* Cardiac insufficiency (NYHA≥ 2)
* Renal insufficiency (GFR ≤ 60 ml/min)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Body composition, especially Extracellular Volume, Intracellular Volume, Total Body Fluid Volume and Fluid Overload. | 6 hours
  The primary outcome parameter is the correct detection of the iv fluid therapy by a corresponding increase in the parameters ExtraCellular Volume (ECV), Total Body Fluid Volume (TBV) and Fluid Overload (FO).

SECONDARY OUTCOMES:
Change over time of the body fluid compartments after iv fluid therapy | 6 hours
  Secondary outcome parameters include the change over time of ICV, ECV, TBV and FO after the iv therapy at the intervention "Fuid Therapy".

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria